CLINICAL TRIAL: NCT05157555
Title: Quality of Life in Patients After Pharyngolaryngectomy
Acronym: LARYNG-QDV
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Université de Reims Champagne-Ardenne (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-010-LARYNG-QDV
Record Dates: First submitted 2021-12-01; First posted 2021-12-15 (Actual); Last update posted 2022-03-25 (Actual); Status verified 2021-12

CONDITIONS: Laryngectomy; Status
Keywords: Laryngeal cancer - laryngectomy - quality of life
MeSH Terms: interventions — Data Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 5 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- "with laryngectomy" group: "with laryngectomy" group: patients with laryngectomy for any type of cancer
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — Description: quality of life assessment

SUMMARY:
Laryngeal cancer is an indication for a laryngectomy (separation of the airways and digestive tract). Laryngectomy causes a permanent disruption of self-perception. Communication, social interactions, diet andaesthetic appearance are altered. Its modifications disrupt the quality of life of patients and must be taken into account as soon as possible in patient cares.

DETAILED DESCRIPTION:
The aim of the study is to describe quality of life in patients with laryngectomy.

ELIGIBILITY:
Inclusion Criteria:

* male or female
* with laryngectomy
* agreeing to participate in the study

Exclusion Criteria:

- less than 18 years old

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients with laryngectomy
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-02-10 (Actual); Primary Completion 2022-05-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
EORTC QLQ-C30 | Day 0
  The QLQ-C30 is a generic questionnaire with 30 questions coded in 4 response modalities (not at all (1), a little (2), enough (3), a lot (4)) or in 7 response modalities (from very bad (1) to excellent ( 7)).
  Questions are summarized in five multiitem domains (physical, role, cognitive, emotional, and social functioning) and nine single item domains (fatigue, pain, nausea/vomiting, appetite loss, financial impact; diarrhea, constipation, sleep disturbance and quality of life).
  Each domain is scored between 0 and 100. For functional domains, a high score value represents a high level of quality of life. For symptom domains, a high score represents an important level of symptoms (a low level of quality of life).

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Gustave Roussy, Villejuif, France

IPD SHARING:
Plan to Share IPD: No